CLINICAL TRIAL: NCT00554008
Title: Randomized, Prospective, Single Blinded Trial of Laparoscopic Versus Open Appendectomy in Children
Brief Title: Comparative Study of Laparoscopic Versus Open Appendectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, David Bliss, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00002184
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Appendicitis
Keywords: Appendicitis; laparoscopy; randomized trial; children; pediatric
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): children randomized to open appendectomy
  Interventions: Procedure: open appendectomy
- 2 (Active Comparator): children randomized to laparoscopic appendectomy
  Interventions: Procedure: laparoscopic appendectomy

INTERVENTIONS:
Procedure: laparoscopic appendectomy — appendix removal via scope
  Arms: 2
Procedure: open appendectomy — open operation for removal of appendix
  Arms: 1

SUMMARY:
The study intends to compare the results of two surgical methods to remove the appendix in children with appendicitis. Specifically, up to 500 children over 3 years will be placed in two groups where the only difference in treatment is open or laparoscopic (scope) operation. Each group will be tracked for their baseline characteristics, events during operation and recovery, pain medication requirements, duration of hospital stay, and patient/family satisfaction.

The investigators hypothesize that their will be no difference in the parameters measured between the techniques of appendix removal.

ELIGIBILITY:
Inclusion Criteria:

* All children under the age of 18 years with diagnosed appendicitis

Exclusion Criteria:

* Refusal of consent
* Primary language other than English or Spanish.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Surgical complications, length of stay, pain medication requirements | within 30 days of intervention

SECONDARY OUTCOMES:
Patient/family satisfaction | within 7 days of intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Bliss, M.D., Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon